CLINICAL TRIAL: NCT04870099
Title: Leveraging Computational Social Sciences and Natural Language Processing to Optimize Engagement and Response to Low-intensity CBT for Depression and Anxiety
Brief Title: Guided Self-help for Common Mental Disorders
Acronym: DWM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana Clinical and Translational Sciences Institute (Other); National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Lorenzo Lorenzo-Luaces, Assistant Professor Pyschological and Brain Sciences, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004321422; KL2TR002530 (NIH); UL1TR002529 (NIH)
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Bibliotherapy

STUDY DESIGN:
Intervention Model Description: Guided self-help
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Guided self-help (Experimental): Participants are given access to the World Health Organization's (WHO) "Doing what matters in times of stress: An illustrated guide" (https://www.who.int/publications/i/item/9789240003927) virtually (i.e., as a pdf) and/or in print. Each participant is assigned an "eCoach" -- an undergraduate, post-baccalaureate, or graduate research assistant -- who will meet with the participant for a 60-minute welcome call describing the intervention and 3-6 sessions of guidance focused on promoting adherence to the manual and using skills in everyday life.
  Interventions: Behavioral: Doing What Matters in Times of Stress: An Illustrated Guide

INTERVENTIONS:
Behavioral: Doing What Matters in Times of Stress: An Illustrated Guide — From the WHO's website: Doing What Matters in Times of Stress: An Illustrated Guide is a stress management guide for coping with adversity. The guide aims to equip people with practical skills to help cope with stress. A few minutes each day are enough to practice the self-help techniques. The guide can be used alone or with the accompanying audio exercises.
  Informed by evidence and extensive field testing, the guide is for anyone who experiences stress, wherever they live and whatever their circumstances.

SUMMARY:
Common mental disorders (CMDs) like depression and anxiety account for a large proportion of disability worldwide. Access to effective treatments like cognitive-behavioral therapy (CBT) is limited and has not reduced the public health burden of psychopathology. For patients with mild-moderate CMDs, lower-intensity treatments like guided self-help CBT (GSH-CBT) are effective and more scalable (e.g., via the internet). The advent of social media has opened avenues for dissemination of GSH-CBTs and allows for passive sensing of mood, thinking, behavior, and social networks. We propose to leverage a social media platform used by over a fifth of the United States (Twitter) as a recruitment tool to virtually screen over 150 individuals, recruit N=60 to a 5-week course of GSH-CBT, and extract social media data from individuals engaged in GSH-CBT. Sociodemographic and social media data will be used to predict engagement, outcomes, and processes in GSH-CBT.

ELIGIBILITY:
Inclusion Criteria:

* At least mild distress: K6 score ≥ 6
* Having reasonably regular access to the internet or a telephone

Exclusion Criteria:

- Suicidality: Patient Health Questionnaire-9 (PHQ9) item 9 ("thoughts that you would be better off dead, or of hurting yourself ") ≥ 2 ("more than half the days")

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Guided Self-help: Participants are given access to the World Health Organization's (WHO) "Doing what matters in times of stress: An illustrated guide" (https://www.who.int/publications/i/item/9789240003927) virtually (i.e., as a pdf) and/or in print. Each participant is assigned an "eCoach" -- an undergraduate, post-baccalaureate, or graduate research assistant -- who will meet with the participant for a 60-minute welcome call describing the intervention and 3-6 sessions of guidance focused on promoting adherence to the manual and using skills in everyday life.
  Doing What Matters in Times of Stress: An Illustrated Guide: From the WHO's website: Doing What Matters in Times of Stress: An Illustrated Guide is a stress management guide for coping with adversity. The guide aims to equip people with practical skills to help cope with stress. A few minutes each day are enough to practice the self-help techniques. The guide can be used alone or with the accompanying audio exercises.
  Informed by evidence and extensive field testing, the guide is for anyone who experiences stress, wherever they live and whatever their circumstances.
Period: Overall Study
Arm/Group | Guided Self-help
Started | 141 (Of these 141 people, 119 actually started the guided self-help (GSH) cognitive-behavioral therapy (CBT))
Completed | 97
Not Completed | 44

BASELINE CHARACTERISTICS:
Population: 141 individuals qualified for the study and reached the onboarding call.
Arm/Group | Guided Self-help
Number analyzed (Participants) | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.36 (13.95)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender identity: Men | 18
  Gender identity: Women | 120
  Gender identity: Genderqueer or non-binary | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Non-Hispanic White | 110
  Race/ethnicity: Non-Hispanic Black | 5
  Race/ethnicity: Hispanic | 11
  Race/ethnicity: Asian | 8
  Race/ethnicity: Other (e.g., multiracial) | 7
Kessler Psychological Distress 6 Scale (K6) [Mean (Standard Deviation); unit: units on a scale] | 10.99 (3.59)

OUTCOME MEASURES:

1. Primary Outcome: 6-week Change in Kessler 6 Psychological Distress Scale (K6)
Description: Changes in K6 from baseline to Week 6. The K6 is a measure of distress and the measure is scored on a scale of 0 - 24 where higher scores indicate higher distress (i.e., are negative). Thus, lower scores relative to baseline indicate more positive outcomes.
Time Frame: Change from Baseline to Week 6
Population: Note: These analyses use imputed data.
Measure: Mean (Standard Deviation); unit: score on a scale (K6)
Arm/Group | Guided Self-help
Number analyzed (Participants) | 141
score on a scale (K6) | -5.68 (3.61)

2. Primary Outcome: 6-week Change in the WHO 5 Well-being Index (WHO-5)
Description: Changes in WHO-5 from baseline to Week 6. The WHO-5 is a measure of well-being and the measure is scored on a scale of 0 - 100 where higher scores indicate higher satisfaction with life (i.e., are positive). Thus, higher scores relative to baseline indicate more positive outcomes.
Time Frame: Change from Baseline to Week 6
Population: Note: These analyses use imputed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Guided Self-help
Number analyzed (Participants) | 141
score on a scale | 13.61 (18.20)

3. Secondary Outcome: 6-week Change in Emotion Regulation Scale (ERQ) - Reappraisal Subscale
Description: Changes in the ERQ Reappraisal subscale from baseline to Week 6. The Reappraisal scale is a measure of regulating emotions by engaging in reappraisal (i.e., changing the one one thinks about an emotion evoking stimuli), widely considered an adaptive strategy. The measured is scored on a 1-7 scale where higher scores indicate greater use of adaptive emotion regulation strategies (i.e., positive). Thus, higher scores relative to baseline indicate more positive outcomes.
Time Frame: Change from Baseline to Week 6
Population: Note: These analyses use imputed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Guided Self-help
Number analyzed (Participants) | 141
score on a scale | 0.89 (1.10)

4. Secondary Outcome: 6-week Change in the Emotion Regulation Scale (ERQ) - Suppression Subscale
Description: Changes in the ERQ Suppression Scale from baseline to Week 6. The ERQ Suppression scale is a measure of regulating emotions by engaging in suppression (i.e., trying not to think or feel), which is considered a maldaptive emotion regulation strategy. The measure is scored on a scale of 1 - 7 where higher scores indicate higher use of suppression (i.e., negative). Thus, lower scores relative to baseline indicate more positive outcomes.
Time Frame: Change from Baseline to Week 6
Population: Note: These analyses use imputed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Guided Self-help
Number analyzed (Participants) | 141
score on a scale | -0.46 (1.18)

5. Secondary Outcome: 3-month Change in Kessler 6 Psychological Distress Scale (K6; 0 - 24)
Description: Changes in K6 from baseline to 3 months after the termination of the study. The K6 is a measure of distress and the measure is scored on a scale of 0 - 24 where higher scores indicate higher distress (i.e., negative). Thus, lower scores relative to baseline indicate more positive outcomes.
Time Frame: Change from Baseline to 3 Months post-treatment
Population: Note: These analyses use imputed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Guided Self-help
Number analyzed (Participants) | 141
score on a scale | -4.91 (3.85)

6. Secondary Outcome: 3-month Change in the WHO 5 Well-being Index (WHO-5)
Description: Changes in WHO-5 from baseline to 3 months after the termination of the study. The WHO-5 is a measure of well-being and the measure is scored on a scale of 0 - 100 where higher scores indicate higher satisfaction with life (i.e., are positive). Thus, higher scores relative to baseline indicate more positive outcomes.
Time Frame: Change from Baseline to 3 Months post-treatment
Population: Note: These analyses use imputed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Guided Self-help
Number analyzed (Participants) | 141
score on a scale | 15.95 (17.32)

ADVERSE EVENTS:
Time Frame: 6-week assessment period
Description: The adverse events we tracked systematically was withdrawal from the study which was operationalized in two different ways including: completing at least 50% of the scheduled GSH-CBT sessions and completing the post-treatment study follow-up.
Arm/Group | Guided Self-help
All-Cause Mortality (participants affected / at risk) | 0/141
Serious Adverse Events (participants affected / at risk) | 0/141
Other Adverse Events (participants affected / at risk) | 44/141
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guided Self-help (N=141)
Study non-engagement (Psychiatric disorders) | 41 (41) — Did the participant fail to complete at least 50% of scheduled assessments?
Study non-response (Psychiatric disorders) | 44 (44) — Did the participant fail to complete the last study assessment?

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-10-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT04870099/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT04870099/SAP_001.pdf
  • Informed Consent Form (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT04870099/ICF_002.pdf